CLINICAL TRIAL: NCT00095121
Title: A Phase 3, Double-Blind, Randomized, Placebo-Controlled Study of the Safety and Efficacy of Adefovir Dipivoxil in Children and Adolescents (Age 2 to Less Than 18) With Chronic Hepatitis B
Brief Title: Safety and Efficacy of Adefovir Dipivoxil in Children and Adolescents With Chronic Hepatitis B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GS-US-103-0518
Record Dates: First submitted 2004-10-29; First posted 2004-11-01 (Estimated); Results first posted 2011-06-03 (Estimated); Last update posted 2012-05-22 (Estimated); Status verified 2012-05

CONDITIONS: Chronic Hepatitis B
Keywords: Hepatitis B; Children; Pediatric; Adefovir Dipivoxil
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — adefovir dipivoxil; Lamivudine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Placebo (PLB) (Placebo Comparator): Participants randomized to receive placebo received placebo during the first 48 weeks of treatment (double-blind phase) and then all eligible participants were administered open-label ADV for the remainder of the study.
  Interventions: Drug: Placebo (PLB); Drug: Lamivudine
- Adefovir Dipivoxil (ADV) (Experimental): Participants randomized to receive ADV received ADV during the first 48 weeks of treatment (double-blind phase) and then all eligible participants were administered open-label ADV for the remainder of the study.
  Interventions: Drug: Adefovir Dipivoxil (ADV); Drug: Lamivudine

INTERVENTIONS:
Drug: Placebo (PLB) — Matching placebo
  Arms: Placebo (PLB)
Drug: Adefovir Dipivoxil (ADV) — 10-mg tablet or 2-mg/mL oral suspension
  Arms: Adefovir Dipivoxil (ADV)
Drug: Lamivudine — 100-mg tablet administered according to package labeling. Lamivudine was to be added to the open-label ADV regimen of subjects with a serum HBV DNA concentration >= 1000 copies/mL at 2 consecutive study visits at or after Study Week 96. If the HBV DNA concentration remained >= 1000 copies/mL at 2 consecutive study visits after the addition of lamivudine, the investigator was required to discontinue all study drugs, perform the early termination ssessments, and have the subject return every 4 weeks for 16 weeks of posttreatment evaluations.

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of adefovir dipivoxil for the treatment of chronic hepatitis B in children and adolescents (age 2 to less than 18 years) following 48 weeks of placebo-controlled, double-blind treatment and following an additional 192 weeks of open-label adefovir dipivoxil treatment.

DETAILED DESCRIPTION:
Weeks 1 through 48 (Study Year 1): The first 48 weeks of the study were a randomized, double-blind, placebo-controlled, parallel-group treatment period. Participants were randomly assigned to treatment in a 2:1 fashion to ADV or PLB. Prior to randomization, eligible participants were classified into 1 of 6 strata based upon age at screening (2 to < 7 years; >= 7 to < 12 years; >= 12 to < 18 years) and prior exposure to treatment for chronic hepatitis B (CHB) (prior treatment; no prior treatment).

Weeks 49 through 240 (Study Years 2 through 5): At Week 48, all placebo-treated participants who did not exhibit HBeAg or hepatitis B surface antigen (HBsAg) seroconversion at Week 44, plus all ADV-treated participants, were offered the opportunity to receive open-label ADV for up to an additional 192 weeks. Any participant with HBV DNA >= 1000 copies/mL at 2 consecutive visits 12 weeks apart was to be discontinued from open-label study treatment. The only exception was for participants in the adolescent age range with prior lamivudine experience who were allowed the opportunity to add lamivudine to ADV; similarly, if combination failed to impart suppression of HBV DNA below 1000 copies/mL (confirmed) discontinuation was necessary. All participants who discontinued study drug due to confirmed seroconversion were requested to continue to return for study visits for the remainder of the study in order to evaluate the durability of seroconversion. Participants who wished to discontinue study treatment and withdraw from the study prior to study completion were requested to return every 4 weeks for 16 weeks for posttreatment evaluations following an early termination visit. Any participants who experienced posttreatment hepatic flares during the 16-week follow-up period were to be followed every 4 weeks until their ALT levels returned to <= 2 times the upper limit of normal (ULN) for a maximum off-treatment follow-up of 6 months. Participants who experienced a severe hepatic flare (per protocol definition) after discontinuation of ADV during the open-label treatment period may have been eligible to receive ADV for treatment of the hepatic flare (after consultation with the Gilead medical monitor).

ELIGIBILITY:
Key Inclusion Criteria:

* Positive HBsAg >= 6 months prior to randomization and positive HBeAg at screening.
* Serum HBV DNA greater than or equal to 1 x 100,000 copies/mL (PCR assay) at initial or confirmatory screening visit.
* Serum ALT levels greater than or equal to 1.5 x ULN at both initial and confirmatory screening visits.
* Compensated liver disease with anticipated survival greater than 12 months and with the following laboratory and clinical parameters within 4 weeks of baseline: *Prothrombin time less than or equal to 1 second above normal range. *Total bilirubin less than 1.3 mg/dL or normal direct bilirubin. *Serum albumin greater than 3 g/dL (greater than 30 g/L). *No clinical history of ascites, variceal bleeding, encephalopathy or splenomegaly. *Adequate renal function defined as creatinine clearance greater than or equal to 80 mL/min (calculated using Schwartz Formula).

Key Exclusion Criteria:

* Received immunoglobulin, interferon or lamivudine therapy within 6 months prior to initial screening visit.
* Participated in any investigational trial with any investigational compound within 2 months prior to initial screening.
* Organ or bone marrow transplant recipients.
* Clinical evidence of decompensated liver disease.
* A Child-Pugh-Turcotte score greater than 6.
* Inability to comply with study requirements.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 173 (Actual)
Dates: Start 2004-06; Primary Completion 2006-05 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Flaherty, PharmD, Study Director — Gilead Sciences
Locations (1):
- Boston, Massachusetts, United States

REFERENCES:
- [Background] Sokal, E, Kelly, D, et al. The Pharmacokinetics (PK) and Safety of a Single Dose of Adefovir Dipivoxil (ADV) in Children and Adolescents (Aged 2-17) with Chronic Hepatitis B. JHepatol,Vol 40(Suppl 1), P. 132, 2004.
- See also: Related Info — http://www.gilead.com
- See also: Study Results — http://www.gileadclinicaltrials.com/pdf/GS-US-103-0518_48wk_synopsis.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant screened on 17 May 2004; first participant randomized on 21 June 2004. Participants from Gilead pharmacokinetics Study GS-02-517 were allowed to enroll regardless of screening serum hepatitis B virus (HBV) deoxyribonucleic acid (DNA) or alanine aminotransferase (ALT) concentration if they met all other entry criteria.
Groups:
- ADV - ADV: Once daily treatment: children aged 2 to <7 years received 0.3 mg/kg oral suspension; children aged >=7 to <12 years received 0.25 mg/kg oral suspension; children aged >=12 to <18 years received 10 mg tablet. The adefovir dipivoxil (ADV) baseline was defined as the day of first dose of ADV (ie, Week 0 for participants originally randomized to double-blind [DB] ADV [ADV-ADV group]). Additionally, ADV week was defined as the windowed visit week relative to ADV baseline. Thus, participants in the ADV-ADV group could have received up to 240 weeks of ADV treatment (ADV Week 240). Lamivudine was to be added to the open-label ADV regimen of subjects between 12 and <18 years old who had prior lamivudine exposure and who had a serum HBV DNA concentration >= 1000 copies/mL at 2 consecutive study visits at or after Study Week 96.
- PLB - ADV: Placebo (PLB) was matched to adefovir dipivoxil treatment (oral suspension or tablet) by age group. The ADV baseline was defined as the day of first dose of ADV (ie, Week 48 for those originally randomized to placebo [PLB-ADV group]). Additionally, ADV week was defined as the windowed visit week relative to ADV baseline. Thus, participants in the PLB-ADV group could receive only up to 192 weeks of open-label (OL) ADV treatment (ADV Week 192). Lamivudine was to be added to the open-label ADV regimen of subjects between 12 and <18 years old who had prior lamivudine exposure and who had a serum HBV DNA concentration >= 1000 copies/mL at 2 consecutive study visits at or after Study Week 96.
Period: Double-Blind (Study Weeks 0 Through 48)
Arm/Group | ADV - ADV | PLB - ADV
Started | 115 | 58
Completed | 112 | 58
Not Completed | 3 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Not Compliant | 2 | 0
Period: Open-Label (Study Weeks 49 Through 240)
Arm/Group | ADV - ADV | PLB - ADV
Started | 108 | 54
Received Lamivudine (LAM) After Week 96 | 21 | 11
Completed | 46 (Completed the 240-week study period either on or off treatment at Week 240.) | 35 (Completed the 240-week study period either on or off treatment at Week 240.)
Not Completed | 62 | 19

BASELINE CHARACTERISTICS:
Groups:
- ADV - ADV: Once daily treatment: children aged 2 to <7 years received 0.3 mg/kg oral suspension; children aged >=7 to <12 years received 0.25 mg/kg oral suspension; children aged >=12 to <18 years received 10 mg tablet. The ADV baseline was defined as the day of first dose of ADV (ie, Week 0 for participants originally randomized to DB ADV [ADV-ADV group]). Additionally, ADV week was defined as the windowed visit week relative to ADV baseline. Thus, participants in the ADV-ADV group could have received up to 240 weeks of ADV treatment (ADV Week 240).
- PLB - ADV: Placebo was matched to adefovir dipivoxil treatment (oral suspension or tablet) by age group. The ADV baseline was defined as the day of first dose of ADV (ie, Week 48 for those originally randomized to placebo [PLB-ADV group]). Additionally, ADV week was defined as the windowed visit week relative to ADV baseline. Thus, participants in the PLB-ADV group could receive only up to 192 weeks of ADV treatment (ADV Week 192).
- Total: Total of all reporting groups
Arm/Group | ADV - ADV | PLB - ADV | Total
Number analyzed (Participants) | 115 | 58 | 173
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 115 | 58 | 173
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 10.8 (4.33) | 10.7 (3.94) | 10.8 (4.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 19 | 60
  Male | 74 | 39 | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 114 | 58 | 172
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 29 | 12 | 41
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 3 | 14
  White | 70 | 41 | 111
  More than one race | 4 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 35 | 13 | 48
  Belgium | 6 | 3 | 9
  Germany | 11 | 8 | 19
  Poland | 48 | 27 | 75
  Spain | 4 | 4 | 8
  United Kingdom | 11 | 3 | 14
Body Mass Index (Males) [Mean (Standard Deviation); unit: kg/cm^2] | 19.3 (4.04) | 19.7 (4.87) | 19.4 (4.33)
Body Mass Index (Females) [Mean (Standard Deviation); unit: kg/cm^2] | 17.8 (3.68) | 17.7 (3.76) | 17.7 (3.67)
Prior Exposure to Hepatitis B Treatment [Number; unit: participants]
  Yes | 64 | 33 | 97
  No | 51 | 25 | 76
HBV DNA [Mean (Standard Deviation); unit: log10 copies/mL] | 8.74 (0.894) | 8.67 (1.016) | 8.71 (0.935)
Hepatitis B Surface Antigen (HBsAg) [Number; unit: participants]
  Negative | 0 | 0 | 0
  Positive | 115 | 58 | 173
Antibody to HBsAg (HBsAb) [Number; unit: participants]
  Negative | 0 | 0 | 0
  Positive | 0 | 0 | 0
  Not Done | 115 | 58 | 173
Hepatitis B e Antigen (HBeAg) [Number; unit: participants]
  Negative | 2 | 1 | 3
  Positive | 113 | 57 | 170
Antibody to HBeAg (HBeAb) [Number; unit: participants]
  Negative | 0 | 0 | 0
  Positive | 2 | 1 | 3
  Not Done | 113 | 57 | 170
ALT [Mean (Standard Deviation); unit: U/L] | 111 (81.6) | 99 (52.8) | 107 (73.3)
ALT [Number; unit: participants]
  >= Upper Limit of Normal (ULN) | 108 | 56 | 164
  <ULN | 7 | 2 | 9
ALT as Multiple of ULN [Number; unit: participants]
  <=median (2.265) | 57 | 30 | 87
  >median (2.265) | 58 | 28 | 86
ALT Category [Number; unit: participants]
  Alanine aminotransferase <=ULN | 8 | 2 | 10
  ULN <alanine aminotransferase <=2*ULN | 37 | 25 | 62
  2*ULN <alanine aminotransferase <=5*ULN | 52 | 26 | 78
  Alanine aminotransferase >5*ULN | 18 | 5 | 23
ALT (Multiples of ULN) [Mean (Standard Deviation); unit: multiples] | 2.9 (2.03) | 2.6 (1.40) | 2.8 (1.85)
Genotype [Number; unit: participants] — Identification of specific HBV genotype (ie, Genotype A, B, C, D, E, or F).
  participants
    HBV Genotype A | 51 | 32 | 83
    HBV Genotype B | 13 | 5 | 18
    HBV Genotype C | 10 | 4 | 14
    HBV Genotype D | 35 | 14 | 49
    HBV Genotype E | 3 | 2 | 5
    HBV Genotype F | 2 | 0 | 2
    Not Done | 1 | 1 | 2
Time Since HBV Diagnosis [Mean (Standard Deviation); unit: years until enrollment] | 6.8 (4.12) | 6.8 (4.06) | 6.8 (4.09)
Mode of HBV Acquisition [Number; unit: participants]
  Perinatal transmission or within 1st year of life | 47 | 24 | 71
  Unknown | 37 | 21 | 58
  Childhood acquisition after 1st year of life | 19 | 8 | 27
  Transfusion or exposure to infected blood products | 8 | 3 | 11
  Other | 4 | 2 | 6
  Intravenous drug user | 0 | 0 | 0
  Missing | 0 | 0 | 0
  Sexual contact with HBV infected person | 0 | 0 | 0
Symptoms of Acute Hepatitis B [Number; unit: participants] — Symptoms of acute HBV infection include fever, fatigue, loss of appetite, nausea, vomiting, abdominal pain, dark urine, clay-colored bowel movements, joint pain, and jaundice. - cdc.gov [homepage on the Internet]. Atlanta: Centers for Disease Control and Prevention. Hepatitis B Information for Health Professionals; [updated 2011 April 4]. Available from: http://www.cdc.gov/hepatitis/HBV/HBVfaq.htm.
  participants
    Yes | 2 | 2 | 4
    No | 113 | 56 | 169
Hepatitis B Flares (Acute Exacerbation) [Number; unit: participants] — A hepatic flare was defined as a) serum ALT > 2 x study baseline and > 10 x ULN or b) an ALT 1-grade shift or ALT 2 x previous value and total bilirubin > 2.5 mg/dL or change from study baseline in total bilirubin = 1.0 mg/dL or change from study baseline in prothrombin time > 2 seconds or serum albumin < 3.0 g/dL or change from study baseline in serum albumin <= -1.0 g/dL.
  participants
    Yes | 12 | 4 | 16
    No | 103 | 54 | 157
Current Alcohol Consumption [Number; unit: participants]
  Yes | 0 | 0 | 0
  No | 115 | 58 | 173
Any Prior Hepatitis B Medication [Number; unit: participants]
  Yes | 66 | 33 | 99
  No | 49 | 25 | 74
Prior Use of Famciclovir [Number; unit: participants]
  Yes | 0 | 1 | 1
  No | 115 | 57 | 172
Prior Use of Lamivudine [Number; unit: participants]
  Yes | 46 | 23 | 69
  No | 69 | 35 | 104
Prior Use of Interferon Alpha [Number; unit: participants]
  Yes | 52 | 28 | 80
  No | 63 | 30 | 93
Prior Use of ADV [Number; unit: participants]
  Yes | 4 | 4 | 8
  No | 111 | 54 | 165
Prior Use of Other Hepatitis B Medications [Number; unit: participants] — "Other hepatitis B medications" include any medications other than famciclovir, lamivudine, lobucavir, thymosin alpha, ganciclovir, interferon alpha, hepatitis B immune globulin (HBIG), entecavir, clevudine, emtricitabine, and ADV.
  participants
    Yes | 8 | 2 | 10
    No | 107 | 56 | 163

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Serum Hepatitis B Virus (HBV) Deoxyribonucleic Acid (DNA) < 1000 Copies/mL (Polymerase Chain Reaction [PCR]-Based Assay) and Normal Alanine Aminotransferase (ALT) at Week 48 (Missing = Failure)
Description: In the absence of biopsy data from these pediatric participants, this endpoint enables assessments of drug effect on viral replication and the underlying degree of inflammation in the liver.
Time Frame: Week 48
Population: All randomized participants who received >= 1 dose study medication. If either endpoint was missing a Week 48 value, Week 44 value was substituted and used in the combined endpoint. If participant did not have serum HBV DNA value at Weeks 44 and 48 or ALT value at Weeks 44 and 48, then participant was considered a failure for the Week-48 analysis.
Measure: Number; unit: percentage of participants
Groups:
- Adefovir Dipivoxil (ADV): Once daily treatment: children aged 2 to <7 years received 0.3 mg/kg oral suspension; children aged >=7 to <12 years received 0.25 mg/kg oral suspension; children aged >=12 to <18 years received 10 mg tablet.
- Placebo (PLB): Placebo was matched to adefovir dipivoxil treatment (oral suspension or tablet) by age group.
Arm/Group | Adefovir Dipivoxil (ADV) | Placebo (PLB)
Number analyzed (Participants) | 115 | 58
percentage of participants
  Baseline | 0 | 0
  Week 24 | 5 | 0
  Week 48 or End of Double-blind Treatment | 19 | 2
Statistical Analysis 1: Comparison: Adefovir Dipivoxil (ADV) vs Placebo (PLB); After unblinding the results, due to the small number of responders in the placebo group, it was determined that a statistical exact test would be more appropriate in the evaluation of treatment group differences than the originally planned 95% confidence intervals of the difference between the groups. Therefore, the results were analyzed by study visit, and a Fisher exact test was used to evaluate treatment differences between the adefovir dipivoxil and placebo groups; Test type: Superiority or Other; p < 0.001, Fisher Exact — End of double-blind treatment

2. Secondary Outcome: Percentage of Participants With Serum HBV DNA < 1000 Copies/mL (PCR-based Assay) While on Treatment (Missing = Failure) (ADV Baseline)
Description: The ADV baseline was defined as the day of first dose of ADV (ie, Week 0 for participants originally randomized to double-blind ADV [ADV-ADV group] and Week 48 for those originally randomized to placebo [PLB-ADV group]).
Time Frame: ADV baseline
Population: The OL analysis set was used for this endpoint and included any participant who took at least 1 dose of open-label ADV. Participants with missing values were considered as failures rather than excluded.
Measure: Number; unit: percentage of participants
Arm/Group | ADV - ADV | PLB - ADV
Number analyzed (Participants) | 108 | 54
percentage of participants | 0 | 0

3. Secondary Outcome: Percentage of Participants With Serum HBV DNA < 1000 Copies/mL (PCR-based Assay) While on Treatment - Missing = Failure) (ADV Week 192)
Description: Adefovir week was defined as the windowed visit week relative to ADV baseline. Thus, participants in the ADV-ADV group could have received up to 240 weeks of ADV treatment (ADV Week 240), whereas participants in the PLB-ADV group could receive only up to 192 weeks of ADV treatment (ADV Week 192).
Time Frame: ADV Week 192
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | ADV - ADV | PLB - ADV
Number analyzed (Participants) | 108 | 54
percentage of participants | 15 | 15

4. Secondary Outcome: Percentage of Participants With Serum HBV DNA < 1000 Copies/mL (PCR-based Assay) While on Treatment (Missing = Failure) (ADV Week 240)
Time Frame: ADV Week 240
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Groups:
- ADV - ADV: Once daily treatment: children aged 2 to <7 years received 0.3 mg/kg oral suspension; children aged >=7 to <12 years received 0.25 mg/kg oral suspension; children aged >=12 to <18 years received 10 mg tablet. The ADV baseline was defined as the day of first dose of ADV (ie, Week 0 for participants originally randomized to double-blind ADV [ADV-ADV group]). Additionally, ADV week was defined as the windowed visit week relative to ADV baseline. Thus, participants in the ADV-ADV group could have received up to 240 weeks of ADV treatment (ADV Week 240).
Arm/Group | ADV - ADV
Number analyzed (Participants) | 108
percentage of participants | 6

5. Secondary Outcome: Percentage of Participants With Serum HBV DNA < 400 Copies/mL (PCR-based Assay) While on Treatment (Missing = Failure) (ADV Baseline)
Description: as for outcome 2
Time Frame: ADV baseline
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | ADV - ADV | PLB - ADV
Number analyzed (Participants) | 108 | 54
percentage of participants | 0 | 0

6. Secondary Outcome: Percentage of Participants With Serum HBV DNA < 400 Copies/mL (PCR-based Assay) While on Treatment (Missing = Failure) (ADV Week 192)
Description: as for outcome 3
Time Frame: ADV Week 192
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | ADV - ADV | PLB - ADV
Number analyzed (Participants) | 108 | 54
percentage of participants | 11 | 13

7. Secondary Outcome: Percentage of Participants With Serum HBV DNA < 400 Copies/mL (PCR-based Assay) While on Treatment (Missing = Failure) (ADV Week 240)
Time Frame: ADV Week 240
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | ADV - ADV
Number analyzed (Participants) | 108
percentage of participants | 6

8. Secondary Outcome: Adefovir (ADV) Baseline Serum HBV DNA
Description: as for outcome 2
Time Frame: ADV baseline
Population: The OL analysis set included any participant who took at least one dose of open-label ADV. This analysis set was also subdivided based on DB drug, as ADV-ADV or PLB-ADV. Analysis set included only data from participants while on study treatment.
Measure: Mean (Standard Deviation); unit: log10 HBV DNA copies/mL
Groups:
- ADV - ADV: Double-blind once daily ADV treatment: children aged 2 to <7 years received 0.3 mg/kg oral suspension; children aged >=7 to <12 years received 0.25 mg/kg oral suspension; children aged >=12 to <18 years received 10 mg tablet. At Week 48, ADV-treated participants were offered the opportunity to receive open-label ADV for up to an additional 192 weeks (ie, OL Weeks 49 to 240). ADV baseline was defined as the day of first dose of ADV (ie, Week 0 for participants originally randomized to double-blind ADV [ADV-ADV group]). ADV week was defined as the windowed visit week relative to ADV baseline. Thus, participants in the ADV-ADV group could have received up to 240 weeks of ADV treatment (ADV Week 240).
- PLB - ADV: Placebo was matched to ADV treatment (oral suspension or tablet) by age group for the DB treatment period. At Week 48, all placebo-treated participants who did not exhibit HBeAg or HBsAg seroconversion at Week 44 were offered the opportunity to receive OL ADV for up to an additional 192 weeks (ie, enter the OL study period; Weeks 49 to 240).The ADV baseline was defined as the day of first dose of ADV (ie, Week 48 for those originally randomized to placebo [PLB-ADV group]). ADV week was defined as the windowed visit week relative to ADV baseline. Thus, participants in the PLB-ADV group could receive only up to 192 weeks of ADV treatment (ADV Week 192).
Arm/Group | ADV - ADV | PLB - ADV
Number analyzed (Participants) | 108 | 54
log10 HBV DNA copies/mL | 8.76 (0.869) | 8.24 (1.248)

9. Secondary Outcome: Change From ADV Baseline to ADV Week 192 for Serum HBV DNA
Description: as for outcome 3
Time Frame: ADV baseline to ADV 192 weeks
Population: The OL analysis set included any participant who took at least one dose of open-label ADV. This analysis set was subdivided based on DB drug, as ADV-ADV or PLB-ADV. Analysis set included only data from participants while on study treatment.
Measure: Mean (Standard Deviation); unit: log10 HBV DNA copies/mL
Arm/Group | ADV - ADV | PLB - ADV
Number analyzed (Participants) | 17 | 9
log10 HBV DNA copies/mL | -5.89 (1.119) | -5.41 (1.573)

10. Secondary Outcome: Change From ADV Baseline to ADV Week 240 for Serum HBV DNA
Time Frame: ADV baseline to ADV 240 weeks
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: log10 HBV DNA copies/mL
Groups:
- ADV - ADV: Double-blind once daily ADV treatment: children aged 2 to <7 years received 0.3 mg/kg oral suspension; children aged >=7 to <12 years received 0.25 mg/kg oral suspension; children aged >=12 to <18 years received 10 mg tablet. At Week 48, ADV-treated participants were offered the opportunity to receive OL ADV for up to an additional 192 weeks (ie, OL Weeks 49 to 240). ADV baseline was defined as the day of first dose of ADV (ie, Week 0 for participants originally randomized to double-blind ADV [ADV-ADV group]). ADV week was defined as the windowed visit week relative to ADV baseline. Thus, participants in the ADV-ADV group could have received up to 240 weeks of ADV treatment (ADV Week 240).
Arm/Group | ADV - ADV
Number analyzed (Participants) | 7
log10 HBV DNA copies/mL | -5.87 (1.826)

11. Secondary Outcome: ADV Baseline ALT
Description: as for outcome 2
Time Frame: ADV baseline
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | ADV - ADV | PLB - ADV
Number analyzed (Participants) | 108 | 54
U/L | 108.69 (79.069) | 99.81 (97.583)

12. Secondary Outcome: Change From ADV Baseline to ADV Week 192 for ALT
Description: as for outcome 3
Time Frame: ADV baseline to ADV 192 weeks
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | ADV - ADV | PLB - ADV
Number analyzed (Participants) | 17 | 8
U/L | -66.06 (42.655) | -38.88 (33.566)

13. Secondary Outcome: Change From ADV Baseline to ADV Week 240 for ALT
Time Frame: ADV baseline to ADV 240 weeks
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | ADV - ADV
Number analyzed (Participants) | 6
U/L | -64.33 (44.742)

14. Secondary Outcome: Percentage of Participants With Normal ALT at Adefovir Baseline (Missing = Failure)
Description: The ADV baseline was defined as the day of first dose of ADV (ie, Week 0 for participants originally randomized to double-blind ADV [ADV-ADV group] and Week 48 for those originally randomized to placebo [PLB-ADV group]). Normal ALT: 0-1 year old = <=54 U/L; females 1-88 years old and males 1-10 years old = 8-34 U/L; males 10-88 years old = 8-43 U/L.
Time Frame: ADV baseline
Population: The OL analysis set included any participant who took at least one dose of open-label ADV. This analysis set was also subdivided based on DB drug, as ADV-ADV or PLB-ADV. Participants with missing values were considered as failures rather than excluded. Analysis set included only data from participants while on study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | ADV - ADV | PLB - ADV
Number analyzed (Participants) | 108 | 54
percentage of participants | 7 | 15

15. Secondary Outcome: Percentage of Participants With Normal ALT at ADV Week 192 (Missing = Failure)
Description: Adefovir week was defined as the windowed visit week relative to ADV baseline. Thus, participants in the ADV-ADV group could have received up to 240 weeks of ADV treatment (ADV Week 240), whereas participants in the PLB-ADV group could receive only up to 192 weeks of ADV treatment (ADV Week 192). Normal ALT: 0-1 year old = <=54 U/L; females 1-88 years old and males 1-10 years old = 8-34 U/L; males 10-88 years old = 8-43 U/L.
Time Frame: ADV Week 192
Population: The OL analysis set included any participant who took at least one dose of open-label ADV. This analysis set was subdivided based on DB drug, as ADV-ADV or PLB-ADV. Participants with missing values were considered as failures rather than excluded. Analysis set included only data from participants while on study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | ADV - ADV | PLB - ADV
Number analyzed (Participants) | 108 | 54
percentage of participants | 14 | 13

16. Secondary Outcome: Percentage of Participants With Normal ALT at ADV Week 240 (Missing = Failure)
Description: Normal ALT: 0-1 year old = <=54 U/L; females 1-88 years old and males 1-10 years old = 8-34 U/L; males 10-88 years old = 8-43 U/L.
Time Frame: ADV Week 240
Population: as for outcome 15
Measure: Number; unit: percentage of participants
Arm/Group | ADV - ADV
Number analyzed (Participants) | 108
percentage of participants | 5

17. Secondary Outcome: Percentage of Participants With Hepatitis B e Antigen (HBeAg) Loss or Seroconversion by End of Blinded Treatment (Study Week 48; Randomized and Treated Analysis Set)
Description: HBeAg loss is defined for an individual participant as HBeAg+ at ADV baseline and HBeAg- post baseline. HBeAg seroconversion is defined for an individual participant as HBeAg+ at ADV baseline and HBeAg- and hepatitis B e antibody + (anti-HBe+) post baseline.
Time Frame: Study Week 0 to Study Week 48 (double-blind period)
Population: The randomized and treated analysis set included all participants who were randomized into the study and received at least one dose of study medication. For Week 48 data; if Week 48 was missing, Week 44 was carried forward; if Week 44 was missing, missing = failure.
Measure: Number; unit: percentage of participants
Groups:
- Adefovir Dipivoxil (ADV): Once daily treatment during the double-blind treatment period: children aged 2 to <7 years received 0.3 mg/kg oral suspension; children aged >=7 to <12 years received 0.25 mg/kg oral suspension; children aged >=12 to <18 years received 10 mg tablet. Randomized and Treated Analysis Set (RAT) included adverse events that occurred up to the last dose of double-blind treatment + 4 days or if discontinued early, 30 days after last double-blind dose.
- Placebo (PBL): Placebo was matched to adefovir dipivoxil treatment (oral suspension or tablet) by age group for the double-blind treatment period. RAT included adverse events that occurred up to the last dose of double-blind treatment + 4 days or if discontinued early, 30 days after last double-blind dose.
Arm/Group | Adefovir Dipivoxil (ADV) | Placebo (PBL)
Number analyzed (Participants) | 113 | 57
percentage of participants
  HBeAg Loss | 17 | 5
  Seroconversion to Anti-HBe | 16 | 5
Statistical Analysis 1: Comparison: Adefovir Dipivoxil (ADV) vs Placebo (PBL); Test type: Superiority or Other; p = 0.051, Fisher Exact — Comparison of HBeAg Loss
Statistical Analysis 2: Comparison: Adefovir Dipivoxil (ADV) vs Placebo (PBL); Test type: Superiority or Other; p = 0.051, Fisher Exact — Comparison of HBeAg Seroconversion

18. Secondary Outcome: Percentage of Participants With HBeAg Loss or Seroconversion by ADV Week 192 (Open Label Analysis Set, Participants Who Were HBeAg Positive at ADV Baseline; Missing = Excluded)
Description: ADV baseline = 1st ADV-dose day = Week 0 for ADV-ADV group and Week 48 for PLB-ADV group. ADV week = windowed visit week relative to ADV baseline. Thus, participants in the ADV-ADV group could have received up to 240 weeks of ADV treatment (ADV Week 240), whereas participants in the PLB-ADV group could receive only up to 192 weeks of ADV treatment (ADV Week 192). HBeAg loss is defined per individual participant as HBeAg+ at ADV baseline and HBeAg- post baseline. HBeAg seroconversion is defined for an individual participant as HBeAg+ at ADV baseline and HBeAg- and anti-HBe+ post baseline.
Time Frame: ADV baseline to ADV Week 192
Population: The OL analysis set included any participant who took at least one dose of open-label ADV. This analysis set was subdivided based on DB drug, as ADV-ADV or PLB-ADV. Participants with missing values were excluded. Analysis set included only data from participants while on study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | ADV - ADV | PLB - ADV
Number analyzed (Participants) | 16 | 9
percentage of participants
  HBeAg Loss | 56 | 33
  Seroconversion to Anti-HBe | 44 | 11

19. Secondary Outcome: Percentage of Participants With HBeAg Loss or Seroconversion by ADV Week 240 (Open Label Analysis Set, Participants Who Were HBeAg Positive at ADV Baseline; Missing = Excluded)
Description: Per protocol, participants could discontinue study medication due to HBeAg seroconversion and remain in the study in order to evaluate the durability of seroconversion. HBeAg loss is defined for an individual participant as HBeAg+ at ADV baseline and HBeAg- post baseline. HBeAg seroconversion is defined for an individual participant as HBeAg+ at ADV baseline and HBeAg- and anti-HBe+ post baseline.
Time Frame: ADV baseline to ADV Week 240
Population: as for outcome 18
Measure: Number; unit: percentage of participants
Arm/Group | ADV - ADV
Number analyzed (Participants) | 6
percentage of participants
  HBeAg Loss | 33
  Seroconversion to Anti-HBe | 17

20. Secondary Outcome: Cumulative Summary of Participants With HBV Genotypic Changes From Baseline (Resistance Surveillance)
Description: Resistance surveillance was conducted annually for all participants who remained on treatment and had HBV DNA concentrations greater than or equal to the level of detection (>= 169 copies/mL) by PCR. The last on-ADV sample for all participants in the study was analyzed in the cumulative Week 240 resistance surveillance analysis.
Time Frame: 240 weeks
Population: Last on-ADV sample through Week 240 was analyzed, and participant was excluded from the cumulative Week 240 analysis if HBV DNA value was < 169 copies/mL at Week 240/last time point or if participant discontinued study drug but remained in study. One ADV-ADV participant had an ADV-specific, conserved-site mutation and is counted twice in the table.
Measure: Number; unit: Participants
Arm/Group | ADV - ADV | PLB - ADV
Number analyzed (Participants) | 74 | 37
Participants
  No genotypic changes from baseline | 48 | 18
  Polymorphic site changes | 17 | 12
  Changes at conserved sites in HBV polymerase | 3 | 3
  Developed mutations specific to ADV/lamivudine | 1 | 0
  Unable to be genotyped | 6 | 4

21. Secondary Outcome: Cumulative Summary of Participants With HBV Genotypic Changes From Baseline (Resistance Surveillance) for Subjects Who Received Combination ADV + Lamivudine Therapy
Description: Resistance surveillance was conducted at Week 240/last on-treatment study visit for all participants who had HBV DNA concentrations greater than or equal to the level of detection (>= 169 copies/mL) by PCR while on combination ADV + lamivudine treatment.
Time Frame: 240 weeks
Population: 32/173 added lamivudine from Weeks 108 - 144. Last on-ADV sample through Week 240 analyzed; participant omitted from cumulative Week 240 analysis if HBV DNA <169 copies/mL at Week 240/last time point or stopped study drug but remained in study. 2 ADV-ADV participants had ADV/lamivudine-specific, conserved-site mutation, and counted 2x in table.
Measure: Number; unit: Participants
Arm/Group | ADV - ADV | PLB - ADV
Number analyzed (Participants) | 14 | 3
Participants
  No genotypic changes from baseline | 5 | 1
  Polymorphic site changes | 3 | 1
  Changes at conserved sites in HBV polymerase | 3 | 1
  Developed mutations specific to ADV and/or LAM | 2 | 0
  Unable to be genotyped | 3 | 0

22. Secondary Outcome: Percentage of Participants With Durable HBeAg Seroconversion
Description: A participant was defined to have durable HBeAg seroconversion only if she/he remained in a seroconverted state (HBeAg-, hepatitis B e antibody + [anti-HBe+]) from the date that she/he first seroconverted through and including her/his last study visit. This endpoint could only be assessed for participants who (HBeAg-) seroconverted on-treatment and subsequently discontinued open-label dosing.
Time Frame: 240 weeks
Population: Participants who discontinued treatment because of confirmed HBeAg seroconversion in Weeks 49 to 240 were to remain in the study through Week 240 to monitor the durability of seroconversion. Any participant who formally stopped drug early and restarted, by definition, did not have durable HBeAg seroconversion.
Measure: Number; unit: Percentage of participants
Arm/Group | ADV - ADV | PLB - ADV
Number analyzed (Participants) | 45 | 24
Percentage of participants | 82 | 71

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the entire 240-week duration of the study (ie, during the 48 weeks of randomized treatment and subsequent 192 weeks of open-label treatment).
Description: Treatment-emergent AEs included AEs collected from the date of the first dose of study drug up to the last day on study (including the follow-up, off study medication period of the study). For those participants who did not enter open-label treatment, AEs were collected until 30 days after last double-blind dose. Only on-treatment AEs are shown.
Groups:
- ADV (Double-Blind): Once daily treatment during the DB treatment period: children aged 2 to <7 years received 0.3 mg/kg oral suspension; children aged >=7 to <12 years received 0.25 mg/kg oral suspension; children aged >=12 to <18 years received 10 mg tablet. Treatment-emergent adverse events (AEs) for the DB period are events that occurred up to the last dose of DB treatment + 4 days or if discontinued early, 30 days after last DB dose.
- PLB (Double-Blind): Placebo was matched to adefovir dipivoxil treatment (oral suspension or tablet) by age group for the DB treatment period. Treatment-emergent AEs for the DB period are events that occurred up to the last dose of DB treatment + 4 days or if discontinued early, 30 days after last DB dose.
- ADV - ADV: Double-blind once daily ADV treatment: children aged 2 to <7 years received 0.3 mg/kg oral suspension; children aged >=7 to <12 years received 0.25 mg/kg oral suspension; children aged >=12 to <18 years received 10 mg tablet. At Week 48, ADV-treated participants were offered the opportunity to receive open-label ADV for up to an additional 192 weeks (ie, OL Weeks 49 - 240). ADV baseline was defined as the day of first dose of ADV (ie, Week 0 for participants originally randomized to DB ADV [ADV-ADV group]). ADV week was defined as the windowed visit week relative to ADV baseline. Thus, participants in the ADV-ADV group could have received up to 240 weeks of ADV treatment (ADV Week 240). Treatment-emergent AEs for the OL period are events that began on or after the date of the first dose of OL ADV, and include only new events (ie, events that were never observed during the DB period, or, events observed during the DB period but with greater severity during the OL period).
- PLB - ADV: Placebo was matched to ADV treatment (oral suspension or tablet) by age group for the DB treatment period. At Week 48, all placebo-treated participants who did not exhibit HBeAg or hepatitis B surface antigen seroconversion at Week 44 were offered the opportunity to receive OL ADV for up to an additional 192 weeks (ie, enter the OL study period; Weeks 49 - 240).The ADV baseline was defined as the day of first dose of ADV (ie, Week 48 for those originally randomized to placebo [PLB-ADV group]). ADV week was defined as the windowed visit week relative to ADV baseline. Thus, participants in the PLB-ADV group could receive only up to 192 weeks of ADV treatment (ADV Week 192). Treatment-emergent AEs for the OL period are events that began on or after the date of the first dose of OL ADV, and include only new events (ie, events that were never observed during the DB period, or, events observed during the DB period but with greater severity during the OL period).
Arm/Group | ADV (Double-Blind) | PLB (Double-Blind) | ADV - ADV | PLB - ADV
Serious Adverse Events (participants affected / at risk) | 7/115 | 5/58 | 10/108 | 3/54
Other Adverse Events (participants affected / at risk) | 95/115 | 47/58 | 73/108 | 46/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ADV (Double-Blind) (N=115) | PLB (Double-Blind) (N=58) | ADV - ADV (N=108) | PLB - ADV (N=54)
diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
pyrexia (General disorders) | 2 | 0 | 0 | 0
hepatitis (Hepatobiliary disorders) | 0 | 1 | 1 | 0
gastroenteritis bacterial (Infections and infestations) | 0 | 1 | 0 | 0
pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 1
hepatic enzyme increased (Investigations) | 1 | 0 | 1 | 0
syncope vasovagal (Nervous system disorders) | 1 | 0 | 0 | 0
convulsion (Nervous system disorders) | 0 | 0 | 1 | 0
abnormal behavior (Psychiatric disorders) | 1 | 0 | 0 | 0
depression (Psychiatric disorders) | 0 | 0 | 1 | 1
osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ADV (Double-Blind) (N=115) | PLB (Double-Blind) (N=58) | ADV - ADV (N=108) | PLB - ADV (N=54)
abdominal pain (Gastrointestinal disorders) | 10 | 9 | 9 | 10
diarrhoea (Gastrointestinal disorders) | 7 | 4 | 5 | 3
vomiting (Gastrointestinal disorders) | 4 | 5 | 4 | 2
abdominal pain upper (Gastrointestinal disorders) | 4 | 1 | 4 | 3
toothache (Gastrointestinal disorders) | 1 | 3 | 0 | 0
pyrexia (General disorders) | 14 | 5 | 5 | 3
nasopharyngitis (Infections and infestations) | 30 | 14 | 12 | 8
pharyngitis (Infections and infestations) | 15 | 7 | 14 | 12
upper respiratory tract infection (Infections and infestations) | 13 | 8 | 6 | 4
rhinitis (Infections and infestations) | 5 | 9 | 0 | 0
bronchitis (Infections and infestations) | 8 | 4 | 6 | 4
influenza (Infections and infestations) | 4 | 3 | 2 | 3
gastroenteritis (Infections and infestations) | 1 | 3 | 0 | 0
tonsillitis (Infections and infestations) | 2 | 2 | 4 | 5
otitis media (Infections and infestations) | 2 | 2 | 0 | 3
headache (Nervous system disorders) | 15 | 8 | 11 | 4
cough (Respiratory, thoracic and mediastinal disorders) | 17 | 12 | 6 | 1
pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 4 | 0 | 0
epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 6 | 1
rash (Skin and subcutaneous tissue disorders) | 3 | 3 | 7 | 3
blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication must include results in their entirety and not as individual center data. Results may be published/presented at scientific meetings. All manuscripts/abstracts must be submitted to Gilead prior to submission. Any formal publication of the study in which input of Gilead personnel exceeded that of conventional monitoring will be considered as a joint publication by the investigator and the appropriate Gilead personnel.